CLINICAL TRIAL: NCT02023710
Title: A Randomized Phase II Study Evaluating the Activity of Bevacizumab in Combination With Carboplatin Plus Paclitaxel in Patients With Previously Untreated Advanced Mucosal Melanoma
Brief Title: Bevacizumab Combined With Carboplatin Plus Paclitaxel Chemotherapy to Treat Metastatic Mucosal Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCH-MM-131101
Record Dates: First submitted 2013-12-19; First posted 2013-12-30 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: mucosal melanoma; Bevacizumab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Melanoma | interventions — Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BEV plus Chemotherapy (Experimental): Paclitaxel 175mg/m2, d1; Carboplatin AUC=5, d1; Bevacizumab 5mg/kg, d1、15; 28 days a cycle
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab
- Chemotherapy alone (Active Comparator): Paclitaxel 175mg/m2, d1; Carboplatin AUC=5, d1; 28 days a cycle
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m^2 by IV infusion on the first day of each 4-week cycle (dose was based on patient's weight and could be adjusted for weight change)
  Other Names: Taxel
Drug: Carboplatin — Dose based on patients' creatinine clearance (Calvert formula) and administered by intravenous (IV) infusion on the first day of each 4-week cycle
  Other Names: CBP
Drug: Bevacizumab — 5mg/kg by intravenous (IV) infusion every two weeks of each 4-week cycle (dose was based on patient's weight at screening and remained the same throughout study)
  Other Names: BEV
  Arms: BEV plus Chemotherapy

SUMMARY:
Mucosal melanoma is rare and associated with extremely poor prognosis.No effective treatment for advanced mucosal melanoma patients.Investigators conducted a randomized phase II study in patients with previously untreated metastatic mucosal melanoma to characterize the efficacy and safety of bevacizumab when combined with carboplatin plus paclitaxel.

DETAILED DESCRIPTION:
Mucosal melanoma is rare and associated with extremely poor prognosis.It is the second most common subtype in Asians.No effective treatment for advanced mucosal melanoma patients.Malignant melanoma is a highly vascular tumor in which vascular endothelial growth factor(VEGF) is strongly expressed and seems to play an important role in disease progression.A randomized phase II study evaluated the activity of Bevacizumab in combination with carboplatin plus paclitaxel(CPB arm) in patients with previously untreated advanced melanoma.Overall response rates was 25.5%,median overall survival time(OS) was 12.3 months in the CPB arm. Investigators conducted a randomized phase II study in patients with previously untreated metastatic mucosal melanoma to characterize the efficacy and safety of bevacizumab when combined with carboplatin plus paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed mucosal melanoma with metastases and has no received any systemic treatment.
2. ECOG performance status 0, 1
3. Estimated life expectancy of 12 weeks or greater
4. Age 18 years or older, male or female
5. At least one measurable site (diameter≥1cm) of disease (RECIST 1.1).
6. Adequate organ function
7. Without symptoms of brain metastases and stable in neuro-functions.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Mutations in C-KIT or BRAF-V600E, asked for other target treatments
2. Pregnant or lactation women
3. Acute infections without control.
4. Heart disease history, cardiac function class≥NYHA II.
5. HIV positive or chronic HBV/HCV in active stage.
6. Brain metastases or primary tumor with positive symptoms
7. Need anti-epileptic treatments
8. Organ transplantation history
9. Hemorrhagic tendency or related history
10. Renal dialysis patients
11. Diagnosis of any second malignancy within the last 3 years, except for adequately treated.
12. Current treatment on another clinical trial
13. The other improper situations which investigator judged.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
progress-free survival(PFS) | From randomization up to 144 weeks
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
adverse event(AE) | From randomization up to144 weeks
  Any events,no matter related to interventions,occur during the period from the enrollment to death or 30 days after withdrawal from the trial
Overall Survival(OS) | Up to 144 weeks
  Overall survival was defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Beijing Cancer Hospital, Beijing
  - Yunan Tumor Hospital, Kunming

REFERENCES:
- [Background] Kim KB, Sosman JA, Fruehauf JP, Linette GP, Markovic SN, McDermott DF, Weber JS, Nguyen H, Cheverton P, Chen D, Peterson AC, Carson WE 3rd, O'Day SJ. BEAM: a randomized phase II study evaluating the activity of bevacizumab in combination with carboplatin plus paclitaxel in patients with previously untreated advanced melanoma. J Clin Oncol. 2012 Jan 1;30(1):34-41. doi: 10.1200/JCO.2011.34.6270. Epub 2011 Nov 28. PMID 22124101
- [Background] Chi Z, Li S, Sheng X, Si L, Cui C, Han M, Guo J. Clinical presentation, histology, and prognoses of malignant melanoma in ethnic Chinese: a study of 522 consecutive cases. BMC Cancer. 2011 Feb 25;11:85. doi: 10.1186/1471-2407-11-85. PMID 21349197
- [Background] Lian B, Si L, Cui C, Chi Z, Sheng X, Mao L, Li S, Kong Y, Tang B, Guo J. Phase II randomized trial comparing high-dose IFN-alpha2b with temozolomide plus cisplatin as systemic adjuvant therapy for resected mucosal melanoma. Clin Cancer Res. 2013 Aug 15;19(16):4488-98. doi: 10.1158/1078-0432.CCR-13-0739. Epub 2013 Jul 5. PMID 23833309
- [Derived] Yan X, Sheng X, Chi Z, Si L, Cui C, Kong Y, Tang B, Mao L, Wang X, Lian B, Li S, Bai X, Zhou L, Dai J, Yao H, Guo J. Randomized Phase II Study of Bevacizumab in Combination With Carboplatin Plus Paclitaxel in Patients With Previously Untreated Advanced Mucosal Melanoma. J Clin Oncol. 2021 Mar 10;39(8):881-889. doi: 10.1200/JCO.20.00902. Epub 2021 Jan 14. PMID 33444116